CLINICAL TRIAL: NCT01026103
Title: A Prospective, Single-center Investigation of the Safety and Performance of the Endo GIA™ Stapler With Endo GIA™ Sulu With Tri-Staple™ Technology in a Gastric Bypass Procedure
Brief Title: Tri Staple Technology Stapler Used in Gastric Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AS09004
Record Dates: First submitted 2009-12-03; First posted 2009-12-04 (Estimated); Results first posted 2014-03-14 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-01

CONDITIONS: Sleep Apnea; Hypertension; Hyperlipidemia; Coronary Artery Disease; Gastroesophageal Reflux Disease; Osteoarthritis; Diabetes
Keywords: gastric bypass; Gastric bypass surgery
MeSH Terms: conditions — Sleep Apnea Syndromes; Hypertension; Hyperlipidemias; Coronary Artery Disease; Gastroesophageal Reflux; Osteoarthritis; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tri Staple (Experimental): This is a single arm study.
  Interventions: Device: Tri Staple Technology stapler

INTERVENTIONS:
Device: Tri Staple Technology stapler — This is a single arm study.

SUMMARY:
The objectives of this clinical trial are to assess in a pilot setting the overall performance and safety of the Endo GIA™ Stapler with Endo GIA™ SULU with Tri-Staple™ Technology when used in a gastric bypass procedure.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be 18-65 years of age.
* The patient has a BMI of 40-60 kg/m2, or 35-40 kg/m2 with one or more of following comorbidities: sleep apnea, hypertension, hyperlipidemia, coronary artery disease, gastro esophageal reflux disease, osteoarthritis, and diabetes and eligible for gastric bypass.
* The patient must be willing and able to participate in the study procedures and able to understand and sign the informed consent.

Exclusion Criteria:

* The procedure is needed as revision bariatric surgery or the patient has had prior gastric surgery (nissen fundoplication, hiatal hernia, etc)
* The patient is pregnant.
* The patient has an active or history of, infection at the operative site.
* The patient is unable or unwilling to comply with the study requirements, follow-up schedule, or to give valid informed consent.
* Patient has an abdominal ventral hernia requiring mesh repair
* The patient has a history of clinically significant liver disease
* The patient has a history of drug or alcohol abuse within 2 years of enrollment
* The patient has a history of venous thrombosis or pulmonary embolism
* The patient has a history of coagulopathy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samer G Mattar, MD, Principal Investigator — Indiana University
Locations (1):
- Clarian Bariatric Center/Indiana University, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: thirty patients consented, 1 was excluded by physician for elevated liver function test; 1 was not considered enrolled as subject did not receive study device in error, leaving 28 enrolled subjects.
Groups:
- Tri Staple: This is a single arm study.
  Tri Staple Technology stapler : This is a single arm study.
Period: Overall Study
Arm/Group | Tri Staple
Started | 30
Consented | 30
Completed | 28
Not Completed | 2
Not completed — Physician Decision | 1
Not completed — did not receive study device bc of error | 1

BASELINE CHARACTERISTICS:
Population: 30 patients consented; 1 patient was withdrawn by physician for elevated liver function test. Twenty-nine (29) patients had baseline characteristics but 1 did not receive study device in error leaving 28 patients enrolled.
Arm/Group | Tri Staple
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With an Uneventful Creation of a Functional Staple Line
Time Frame: Day 0
Measure: Number; unit: participants
Arm/Group | Tri Staple
Number analyzed (Participants) | 28
participants | 28 [88 to 100]

2. Secondary Outcome: Incidence of Intra-operative Bleeding Requiring Intervention
Time Frame: Day 0 and 1 month
Measure: Number; unit: participants
Arm/Group | Tri Staple
Number analyzed (Participants) | 28
participants | 19 [48 to 84]

3. Secondary Outcome: Length of Hospital Stay
Time Frame: Date of discharge which averages 3 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tri Staple
Number analyzed (Participants) | 28
days | 3.2 (0.5)

4. Secondary Outcome: Incidence of Serosal Tearing
Time Frame: 30 days post op
Measure: Number; unit: participants
Arm/Group | Tri Staple
Number analyzed (Participants) | 28
participants | 0

ADVERSE EVENTS:
Time Frame: 30 days post surgery
Arm/Group | Tri Staple
Serious Adverse Events (participants affected / at risk) | 2/28
Other Adverse Events (participants affected / at risk) | 24/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tri Staple (N=28)
Stricture (Gastrointestinal disorders) | 2 (2)
GI Bleed (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tri Staple (N=28)
Bloating (Gastrointestinal disorders) | 2 (2)
Blood Loss (Surgical and medical procedures) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Depression (Psychiatric disorders) | 7 (7)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Edema (Skin and subcutaneous tissue disorders) | 3 (3)
Fatigue (General disorders) | 19 (19)
Hypertension (Cardiac disorders) | 2 (2)
Infection (Infections and infestations) | 3 (3)
Nausea (General disorders) | 14 (14)
Pain (Surgical and medical procedures) | 10 (10)
Ulcer (Gastrointestinal disorders) | 2 (2)
Vomitting (General disorders) | 6 (6)
Constipation (Gastrointestinal disorders) | 18 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No